CLINICAL TRIAL: NCT06269016
Title: Effect of Hip Strengthening Exercises and Pelvic Floor Exercises on Stress Urinary Incontinence in Postnatal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Sherif Mohamed Hassan, PhD researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003888
Record Dates: First submitted 2024-01-27; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group no intervention (Experimental): no intervention for 3 months with assessment for maximum vaginal squeeze pre and post experiment using bio feedback device and urinary distress inventory UDI-6 short form.
  Interventions: Other: expremental pre and post test
- study group hip muscles strengthening exercise. (Experimental): hip muscles exercises (hip abductors, adductors and gluteus maximus) for 3 months with assessment for maximum vaginal squeeze pre and post experiment using bio feedback device and urinary distress inventory UDI-6 short form.
  Interventions: Other: expremental pre and post test
- study group hip muscles strengthening exercise combined with pelvic floor muscles exercise. (Experimental): hip muscles exercises (hip abductors, adductors and gluteus maximus) combined with pelvic floor muscles exercises for 3 months with assessment for maximum vaginal squeeze pre and post experiment using bio feedback device and urinary distress inventory UDI-6 short form.
  Interventions: Other: expremental pre and post test
- study group pelvic floor muscles exercise. (Experimental): pelvic floor muscles exercises for 3 months with assessment for maximum vaginal squeeze pre and post experiment using bio feedback device and urinary distress inventory UDI-6 short form.
  Interventions: Other: expremental pre and post test

INTERVENTIONS:
Other: expremental pre and post test — effect of strengthening exercise of combined hip strengthening exercises and pelvic floor exercises

SUMMARY:
this study will investigate effect of hip strengthening exercises and pelvic floor exercises on stress urinary incontinence in postnatal women. Clinical practice guidelines recommend PFMT as the first-line treatment for female SUI . Also, it has been speculated that the hip muscles are involved in the continence mechanism and that their deficiency could destabilize the normal function of the system. The addition of hip muscle exercises, regardless of PFM contractions, aimed to improve muscular condition for the motor or synergic strategies in PFM contraction. Secondary effects of these techniques, such as the influence of passive lumbar rotational mobilization in improving hip flexor strength, have been of high interest in physiotherapy in general

ELIGIBILITY:
Inclusion Criteria:

1. Their ages will be ranged from 30 to 35 years old.
2. Their BMI will not exceed 35 Kg/m2.
3. All patients will be multipara women.
4. Their deliveries were normal vaginal delivery.
5. All patients will be diagnosed by gynecologist as mild or moderate degree of SUI.
6. All patients will have the same medical treatment and free from any pathological conditions that might affect the result.

Exclusion Criteria:

1. Recurrent urinary tract infections.
2. Hypertension.
3. Diabetes mellitus.
4. Intra uterine device.
5. Hysterectomy.

Ages: 30 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — stress urinary incomitance post-natal common problem in multiparas' females due to the effect of pregnancy hormones and increase intra-abdominal pressure during pregnancy also normal vaginal delivery increase the weakness of pelvic floor muscles.
Enrollment: 120 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
hip muscles strengthening exercise. | 3 months
  measure the muscle power and endurance for pelvic floor muscles by using bio feedback device to measure maximum vaginal squeeze

CONTACTS AND LOCATIONS:
Locations (1):
- Mai Mohamed Sherif Mohamed Hassan, Cairo, Egypt